CLINICAL TRIAL: NCT03283371
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study Exploring the Efficacy, Safety, and Tolerability of Natalizumab (BG00002) as Adjunctive Therapy in Adult Subjects With Drug-Resistant Focal Epilepsy
Brief Title: Phase 2 Efficacy, Safety, and Tolerability Study of Natalizumab in Focal Epilepsy
Acronym: OPUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101EP201; 2017-001995-45 (EudraCT Number)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Epilepsy, Focal Seizures, Partial Seizures
Keywords: Drug Resistant Focal Epilepsy, Natalizumab, Seizure
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Natalizumab

STUDY DESIGN:
Intervention Model Description: This is a 6-month randomized, double-blind, placebo-controlled study to assess the efficacy, safety, and tolerability of natalizumab as adjunctive therapy in the treatment of adult subjects with drug-resistant focal epilepsy. The placebo-controlled phase is followed by a 6-month open-label phase during which all subjects receive natalizumab.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Natalizumab 300 mg (Experimental): Participants will undergo a prospective baseline period of 6 weeks (Weeks -6 to 0) followed by placebo controlled phase to receive natalizumab 300 mg intravenous (IV) infusion every 4 weeks from Week 0 to Week 24. Participants will continue to receive natalizumab 300 mg IV infusion every 4 weeks for up to an additional 24 weeks in open label phase.
  Interventions: Drug: Natalizumab
- Placebo (Placebo Comparator): Participants will undergo a prospective baseline period of 6 weeks (Weeks -6 to 0) followed by placebo controlled phase to receive natalizumab matching placebo intravenous (IV) infusion every 4 weeks from Week 0 to Week 24. Participants will then receive natalizumab 300 mg IV infusion every 4 weeks for 24 weeks in open label phase.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Natalizumab — As specified in the treatment arm.
  Other Names: Tysabri
  Arms: Natalizumab 300 mg
Other: Placebo — As specified in treatment arms.
  Arms: Placebo

SUMMARY:
The primary efficacy objective of the study is to determine if adjunctive therapy of natalizumab 300 mg intravenous (IV) every 4 weeks reduces the frequency of seizures in adult participants with drug-resistant focal epilepsy. The secondary efficacy objective is to assess the effects of natalizumab versus placebo in drug-resistant focal epilepsy on additional measures of seizure frequency.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have focal epilepsy diagnosed on clinical grounds and as applicable supported by electroencephalogram findings [Scheffer 2017] and brain imaging. Participants with multifocal epilepsy may be included if all other entry criteria are met.
* Must have a drug-resistant epilepsy defined as failure of adequate trials of 2 (or more) tolerated and appropriately chosen and used AEDs (whether as monotherapies or in combination) [Kwan 2010].
* Experiences 6 or more seizures during the 6-week prospective baseline period and is not seizure free for more than 21 consecutive days during the prospective baseline period

Key Exclusion Criteria:

* Focal aware seizures without motor signs are the only seizure type.
* Diagnosis of generalized, combined generalized and focal, or unknown epilepsy
* Known progressive structural CNS lesion.
* History of seizures occurring in predominantly clustered patterns, as determined by the Investigator, over the 12 months prior to the Screening Visit (Week -6) or during the 6-week prospective baseline period, where individual seizures cannot be counted.
* History of status epilepticus within the previous 6 months.
* Known history or presence of non-epileptic seizures.

NOTE; Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (29):
- United States (29):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Bethesda, Maryland
  - Research Site, Chevy Chase, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Saginaw, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Renton, Washington

REFERENCES:
- [Derived] French JA, Cole AJ, Faught E, Theodore WH, Vezzani A, Liow K, Halford JJ, Armstrong R, Szaflarski JP, Hubbard S, Patel J, Chen K, Feng W, Rizzo M, Elkins J, Knafler G, Parkerson KA; OPUS Study Group. Safety and Efficacy of Natalizumab as Adjunctive Therapy for People With Drug-Resistant Epilepsy: A Phase 2 Study. Neurology. 2021 Nov 2;97(18):e1757-e1767. doi: 10.1212/WNL.0000000000012766. Epub 2021 Sep 14. PMID 34521687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 31 investigational sites in United States from 20 March 2018 to 18 Nov 2020.
Pre-assignment Details: A total 67 participants with drug-resistant focal epilepsy were enrolled and randomized in this study. Of which, 66 participants received at least one dose of study drug.
Groups:
- Placebo (Placebo-controlled Phase): Participants received natalizumab-matching placebo intravenous (IV) infusion every 4 weeks in Placebo-controlled Phase for up to Week 24.
- Natalizumab 300 mg (Placebo-controlled Phase): Participants received natalizumab 300 mg IV infusion every 4 weeks in Placebo-controlled Phase for up to Week 24.
- Placebo to Natalizumab 300 mg (Open-label Phase): Participants who received natalizumab-matching placebo in Placebo-controlled Phase, received natalizumab 300 mg IV infusion every 4 weeks in Open-label Phase for up to Week 48.
- Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase): Participants who received natalizumab 300 mg in Placebo-controlled Phase, continued to receive natalizumab 300 mg IV infusion every 4 weeks in Open-label Phase for up to Week 48.
Period: Placebo-controlled
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase) | Placebo to Natalizumab 300 mg (Open-label Phase) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase)
Started | 34 | 33 | 0 | 0
Number of Participants Dosed | 34 | 32 | 0 | 0
Completed | 31 | 30 | 0 | 0
Not Completed | 3 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Participants Did Not Receive Study Drug | 0 | 1 | 0 | 0
Period: Open-label Phase
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase) | Placebo to Natalizumab 300 mg (Open-label Phase) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase)
Started | 0 | 0 | 31 | 30
Completed | 0 | 0 | 27 | 29
Not Completed | 0 | 0 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) population is defined as all participants who were randomized and received any dose of study treatment. Ethnicity was not collected in this study.
Groups:
- Placebo (Placebo-controlled Phase): Participants received natalizumab-matching placebo IV infusion every 4 weeks in Placebo-controlled Phase for up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase) | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.17) | 42.8 (14.56) | 40.9 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 8 | 7 | 15
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log-Transformed Seizure Frequency During Weeks 8 to 24 of Treatment
Description: Seizures included were focal aware seizures with motor signs, focal impaired awareness seizures and focal to bilateral tonic-clonic seizure. Focal aware seizures without motor signs were not included. Seizure clusters (where individual seizures cannot be distinguished) were counted as 1 seizure per cluster on each day that they are present. Study baseline seizure frequency (number of seizures per 28 days) was calculated based on participant's seizure diary data during prospective baseline phase. Seizure frequency (SF) at post baseline visit was calculated based on sum of the seizures reported in participant seizure diary and the number of days with non-missing SF data in participant seizure diary on or after the previous visit date. Change from Baseline are based on natural log transformation of baseline SF or SF at post baseline visit correspondingly. For log-transformation, the quantity 0.2 {ln(x+0.2)} was added to the SF at post baseline visit to account for 0 seizure count.
Time Frame: Baseline, Week 8 to Week 24
Population: ITT population is defined as all participants who were randomized and received any dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: log(seizure/28 days)
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase)
Number analyzed (Participants) | 34 | 32
log(seizure/28 days) | -0.43 (0.162) | -0.58 (0.165)
Statistical Analysis 1: Comparison: Placebo (Placebo-controlled Phase) vs Natalizumab 300 mg (Placebo-controlled Phase); Analysis is based on MMRM and adjusted for natural log-transformed baseline seizure frequency, high seizure frequency category (>=24 seizures and <24 seizures), structural etiology category (yes and no), visit, treatment and treatment by visit interaction. An unstructured variance-covariance matrix is used in the model; Test type: Superiority; p = 0.5053, Mixed Model for Repeated Measures (MMRM); LS Mean logarithmic difference = -0.16, 95% CI 2-sided [-0.62 to 0.31]

2. Secondary Outcome: Percentage of Responders During Weeks 8 to 24 of Treatment
Description: Responders were defined as participants with >=50% reduction from study baseline in seizure frequency during Weeks 8 to 24. Study baseline seizure frequency (number of seizures per 28 days) was calculated based on participants' seizure diary data during the prospective Baseline Phase (number of seizures during Baseline Phase/number of days with non-missing seizure frequency*28). Participants who withdrew from treatment or required protocol specified modifications of antiepileptic drug (AEDs) prior to Week 24 (completion of the Placebo-controlled Phase) or death related to Epilepsy were considered as non-responders in the analysis. Seizure frequency at post baseline visit was calculated based on the sum of the seizures reported in the subject seizure diary and the number of days with non-missing seizure frequency data in the subject seizure diary on or after the previous visit date.
Time Frame: Week 8 to Week 24
Population: The ITT population is defined as all participants who were randomized and received any dose of study treatment.
Measure: Number; unit: percentage of responders
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase)
Number analyzed (Participants) | 34 | 32
percentage of responders | 17.6 | 31.3
Statistical Analysis 1: Comparison: Placebo (Placebo-controlled Phase) vs Natalizumab 300 mg (Placebo-controlled Phase); Based on logistic regression with a term for treatment group and with adjustment for natural log-transformed baseline seizure frequency, high seizure frequency category (>=24 seizures and <24 seizures) and structural etiology category (yes and no); Test type: Superiority; p = 0.2231, Regression, Logistic; Odds Ratio (OR) = 2.09, 95% CI 2-sided [0.64 to 6.85]

3. Secondary Outcome: Number of Participants Free From Seizures During Weeks 8 to 24 of Treatment
Description: Seizure free is defined as a participant with no seizure reported and no missing diary during Weeks 8 to 24. Participants who withdrew from treatment, required modifications of AEDs prior to Week 24 (completion of the Placebo-controlled Phase), or any missing diary data during Weeks 8 to 24 of treatment were not considered as seizure free in the analysis.
Time Frame: Week 8 to Week 24
Population: The ITT population is defined as all participants who were randomized and received any dose of study treatment. Here, "number of participants analyzed" signifies number of participants who were analyzed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase)
Number analyzed (Participants) | 34 | 31
Participants | 1 | 0

4. Secondary Outcome: Percent Change From Baseline of Seizure-Free Days Change During Weeks 8 to 24 of Treatment
Description: Study baseline seizure free days (number of seizure free days per 28 days) was calculated based on the diary data during the prospective baseline Phase (Number of seizures during baseline Phase/Number of days with non-missing seizure frequency*28). Seizure frequency at post baseline visit was calculated based on the sum of the seizures reported in the subject seizure diary and the number of days with non-missing seizure frequency data in the subject seizure diary on or after the previous visit date.
Time Frame: Baseline, Week 8, Week 12, Week 16, Week 20, Week 24
Population: ITT population is defined as all participants who were randomized and received any dose of study treatment. Here, "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase)
Number analyzed (Participants) | 34 | 32
percent change
  Baseline | 16.23 (7.347) | 17.54 (7.223)
  Week 8: number analyzed (Participants) | 31 | 30
  Week 8 | 4.33 (50.740) | 39.23 (130.988)
  Week 12: number analyzed (Participants) | 31 | 30
  Week 12 | 2.41 (52.613) | 32.59 (104.775)
  Week 16: number analyzed (Participants) | 30 | 30
  Week 16 | -0.40 (43.380) | 44.04 (153.714)
  Week 20: number analyzed (Participants) | 30 | 30
  Week 20 | 18.48 (101.318) | 40.44 (144.768)
  Week 24: number analyzed (Participants) | 29 | 29
  Week 24 | 4.27 (47.125) | 33.92 (114.436)

5. Secondary Outcome: Percentage of Participants With Inadequate Treatment Response During Weeks 8 to 24 of Treatment
Description: Inadequate treatment response includes participants who withdraw from treatment due to lack of efficacy or require protocol specified modifications of antiepileptic drugs (AEDs) prior to Week 24 (completion of the placebo- controlled phase) or death related to Epilepsy.
Time Frame: Week 8 to Week 24
Population: The ITT population is defined as all participants who were randomized and received any dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase)
Number analyzed (Participants) | 34 | 32
percentage of participants | 6 | 3
Statistical Analysis 1: Comparison: Placebo (Placebo-controlled Phase) vs Natalizumab 300 mg (Placebo-controlled Phase); Based on the logistic regression model with a term for treatment group and with adjustment for log-transformed baseline seizure frequency, high seizure frequency category (>=24 seizures and <24 seizures) and structural etiology category (yes and no) are considered as covariates; Test type: Superiority; p = 0.6854, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.10 to 4.57]

6. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, in the view of the Investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a birth defect.
Time Frame: From first dose up to 24 weeks after the last dose of study treatment (up to Week 68)
Population: The safety population is defined as all participants who were randomized and received any dose of study treatment and were used for the analysis of safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase) | Placebo to Natalizumab 300 mg (Open-label Phase) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase)
Number analyzed (Participants) | 34 | 32 | 31 | 30
Participants
  AEs | 22 | 24 | 20 | 17
  SAEs | 1 | 1 | 3 | 2

7. Other Pre Specified Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: The laboratory assessments included hematology, blood chemistry, serology, urinalysis and vital signs assessment.
Time Frame: From first dose up to 16 weeks after the last dose of study treatment (up to Week 60)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase) | Placebo to Natalizumab 300 mg (Open-label Phase) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase)
Number analyzed (Participants) | 34 | 32 | 31 | 30
Participants | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) or C-SSRS Score
Description: C-SSRS is a prospective assessment tool to evaluate suicidal ideation and behavior. C-SSRS score for suicidal ideation ranges from 1 to 10, where 1=Wish to be Dead; 2=Nonspecific Active Suicidal Thoughts; 3=Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; 4=Active Suicidal Ideation with Some Intent to Act, without Specific Plan; 5=Active Suicidal Ideation with Specific Plan and Intent; and for suicidal behavior ranges from 6=Preparatory Acts or Behavior, 7=Aborted Attempt, 8=Interrupted Attempt, 9=Actual Attempt (nonfatal), 10=Completed Suicide. Participants with a C-SSRS score between 1-10 are reported in this outcome measure.
Time Frame: Placebo-controlled Phase: Baseline, Weeks 4, 8, 12, 16, 20 and 24; Open-label Phase: Baseline, Weeks 28, 32, 36, 40, 44, 48 and 60/End of Study (EOS)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo-controlled Phase) | Placebo to Natalizumab 300 mg (Open-label Phase) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase)
Number analyzed (Participants) | 34 | 32 | 31 | 30
Participants
  Baseline: Suicidal Ideation or Behavior (1-10) | 0 | 1 | 1 | 1
  Week 4: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 34 | 32 | 0 | 0
  Week 4: Suicidal Ideation or Behavior (1-10) | 0 | 0 |  |
  Week 8: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 34 | 32 | 0 | 0
  Week 8: Suicidal Ideation or Behavior (1-10) | 0 | 0 |  |
  Week 12: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 34 | 32 | 0 | 0
  Week 12: Suicidal Ideation or Behavior (1-10) | 0 | 1 |  |
  Week 16: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 34 | 32 | 0 | 0
  Week 16: Suicidal Ideation or Behavior (1-10) | 0 | 3 |  |
  Week 20: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 34 | 32 | 0 | 0
  Week 20: Suicidal Ideation or Behavior (1-10) | 1 | 2 |  |
  Week 24: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 34 | 32 | 0 | 0
  Week 24: Suicidal Ideation or Behavior (1-10) | 1 | 2 |  |
  Week 28: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 0 | 0 | 31 | 30
  Week 28: Suicidal Ideation or Behavior (1-10) |  |  | 3 | 2
  Week 32: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 0 | 0 | 31 | 30
  Week 32: Suicidal Ideation or Behavior (1-10) |  |  | 1 | 2
  Week 36: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 0 | 0 | 31 | 30
  Week 36: Suicidal Ideation or Behavior (1-10) |  |  | 1 | 1
  Week 40: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 0 | 0 | 31 | 30
  Week 40: Suicidal Ideation or Behavior (1-10) |  |  | 1 | 2
  Week 44: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 0 | 0 | 31 | 30
  Week 44: Suicidal Ideation or Behavior (1-10) |  |  | 1 | 2
  Week 48: Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 0 | 0 | 31 | 30
  Week 48: Suicidal Ideation or Behavior (1-10) |  |  | 1 | 2
  Week 60/End of Study (EOS): Suicidal Ideation or Behavior (1-10): number analyzed (Participants) | 0 | 0 | 31 | 30
  Week 60/End of Study (EOS): Suicidal Ideation or Behavior (1-10) |  |  | 0 | 2

ADVERSE EVENTS:
Time Frame: From first dose up to 24 weeks after the last dose of study treatment (up to Week 68)
Description: The safety population is defined as all participants who were randomized and received any dose of study treatment and were used for the analysis of safety data.
Groups:
- Natalizumab 300 mg (Placebo- Controlled Phase): Participants received natalizumab 300 mg IV infusion every 4 weeks in Placebo-controlled Phase for up to Week 24.
Arm/Group | Placebo (Placebo-controlled Phase) | Natalizumab 300 mg (Placebo- Controlled Phase) | Placebo to Natalizumab 300 mg (Open-label Phase) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/32 | 3/31 | 2/30
Other Adverse Events (participants affected / at risk) | 15/34 | 17/32 | 13/31 | 9/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo-controlled Phase) (N=34) | Natalizumab 300 mg (Placebo- Controlled Phase) (N=32) | Placebo to Natalizumab 300 mg (Open-label Phase) (N=31) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase) (N=30)
Seizure (Nervous system disorders) | 1 | 1 | 1 | 1
Seizure cluster (Nervous system disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo-controlled Phase) (N=34) | Natalizumab 300 mg (Placebo- Controlled Phase) (N=32) | Placebo to Natalizumab 300 mg (Open-label Phase) (N=31) | Natalizumab 300 mg to Natalizumab 300 mg (Open-label Phase) (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1
Amnesia (Nervous system disorders) | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 1 | 2
Headache (Nervous system disorders) | 5 | 6 | 3 | 3
Somnolence (Nervous system disorders) | 3 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Flushing (Vascular disorders) | 3 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT03283371/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT03283371/SAP_001.pdf